CLINICAL TRIAL: NCT00739609
Title: A Phase I Study of Indoximod [1-methyl-D-tryptophan (D-1MT)] in Patients With Relapsed or Refractory Solid Tumors
Brief Title: IDO Inhibitor Study for Relapsed or Refractory Solid Tumors
Acronym: D-1MT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG2100; NCT00788086 (obsolete NCT alias)
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer; Lung Cancer; Melanoma; Pancreatic Cancer; Solid Tumors
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Melanoma; Pancreatic Neoplasms | interventions — 1-methyltryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: 1-methyl-D-tryptophan

INTERVENTIONS:
Drug: 1-methyl-D-tryptophan — D-1MT will be administered in escalating doses. Initial dosing will be 200 mg by mouth daily with escalation planned to 2000 mg by mouth daily and potentially higher doses in subsequent cohorts if tolerated and pharmacokinetic and biologic data support further dose escalation.
  Other Names: D-1MT, NSC-721782, 1-MT

SUMMARY:
This study provides an early evaluation of an entirely new class of small molecule agents directed at disruption or elimination of tumor tolerance, a phenomenon now demonstrated to be involved in the growth of many solid tumors.

DETAILED DESCRIPTION:
This protocol provides an early evaluation of an entirely new class of small molecule agents directed at disruption or elimination of tumor tolerance, a phenomenon now demonstrated to be involved in the growth of many solid tumors. D-1MT, or any other substance targeting this enzymatic pathway indoleamine-(2,3)-dioxygenase (IDO), has not been used previously in humans. Although pre-clinical toxicology in rats and dogs shows an extremely encouraging toxicity profile, the study needs to carefully evaluate the toxicities and pharmacokinetics to provide the basis for assigning a safe and biologically effective dosing regimen for later trials determining its contribution to tumor responses in phase II and III clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* A histological or cytological diagnosis of recurrent or refractory solid tumor malignancy. The patient's pathology must be reviewed and confirmed prior to enrollment (outside reviews acceptable). If no standard therapy exists for disease or subject refused standard therapy, subject would be considered eligible for enrollment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* Hemoglobin ≥ 9.0 gm/dL, absolute neutrophil count (ANC) ≥1200/mm3, platelets ≥100,000/mm3, absolute lymphocyte count ≥800/mm3.
* Hepatic: serum total bilirubin ≤ 1.5 x ULN mg/dL, ALT (SGPT) and AST (SGOT) ≤2.5 x upper limit of normal (ULN).
* Renal: serum creatinine (sCr) ≤1.5 x ULN, or creatinine clearance (Ccr) ≥50 mL/min (approximation by Cockcroft and Gault accepted)
* Life expectancy of greater than 4 months.
* Measurable or non-measurable disease
* Normal EKG including benign variants or abnormalities associated with any condition currently responding to appropriate care (e.g., controlled hypertension with minimal or moderate LVH, controlled AF).
* Prior therapy may include any number of chemotherapy, immunotherapy, and/or radiation therapy regimens. Major surgery or systemic chemotherapy must have been completed at least 4 weeks prior to enrollment and residual toxicities from that therapy must be Grade 1 or lower at the time of enrollment with the exception of hemoglobin and absolute granulocyte count. Localized radiation therapy must have been completed at least 2 weeks prior to enrollment and residual toxicities must be Grade 1 or lower at the time of enrollment.
* Patients must have the ability to understand the study, its inherent risks, side effects and potential benefits and be able to give written informed consent to participate.
* Male and female subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental drug, and for one month after the last dose of drug.
* Patients must be at least 18 years of age

Exclusion Criteria:

* Active CNS metastases or carcinomatous meningitis. Patients with CNS metastases must be at least 3 months status post of prior therapy to the brain and be off all steroids without progressing CNS disease.
* Pregnant or nursing women due to the unknown effects of study drug on the developing fetus or newborn infant.
* History of gastrointestinal disease causing malabsorption or obstruction such as but not limited to Crohn's disease, celiac sprue, tropical sprue, bacterial overgrowth/blind loop syndrome, gastric bypass surgery, strictures, adhesions, achalasia, bowel obstruction, or extensive small bowel resection.
* History of organ transplant.
* Subjects with autoimmune disease, either active or by history (e.g., systemic lupus erythematosis (SLE), rheumatoid arthritis (RA), scleroderma, dermatomyositis, etc.).
* Subjects receiving immunosuppressive therapy including systemic corticosteroid therapy and/other immunosuppressive therapy (methotrexate, cyclosporine, FK-506, rapamycin) for any reason. Subjects receiving inhaled or topical corticosteroids are eligible.
* Significant or uncontrolled cardiovascular disease to include: uncontrolled hypertension (blood pressure must be ≤ 150/90 mmHg at the time of enrollment on a stable antihypertensive regimen); New York Heart Association grade II or greater congestive heart failure (CHF); grade II or greater peripheral vascular disease; significant ventricular arrhythmias requiring medication; and myocardial infarction or unstable angina < six months prior to enrollment.
* Active uncontrolled infection requiring antibiotics within 1-week prior to study, including unexplained fever (temp > 38.1°C or >100.6°F).
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc.).
* No supplements containing L-trytophan or derivatives thereof are allowed to be taken while on study.
* Patients with positive serology for HIV, Hepatitis B or C, and patients with other acquired/inherited immunodeficiencies are ineligible due to the possibility of affecting the response to D-1MT and the higher risk of active opportunistic infections.
* Patients with more than one active malignancy at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Determine the safety and efficacy of administration of D-1MT into patients with recurrent or refractory solid tumors. Establish the toxicities of D-1MT and define any dose limiting toxicities if they occur below the maximum doses. | 6 months

SECONDARY OUTCOMES:
Preliminarily characterize effects of D-1MT on serum kynurenine levels as a biomarker for systemic IDO activity. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles J. Link, M.D., Study Chair — NewLink Genetics Corporation
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Ino K. Indoleamine 2,3-dioxygenase and immune tolerance in ovarian cancer. Curr Opin Obstet Gynecol. 2011 Feb;23(1):13-8. doi: 10.1097/GCO.0b013e3283409c79. PMID 20930628